CLINICAL TRIAL: NCT05955300
Title: Evidence Based Training Program Combined With Nutrition Therapy for Patients With Knee Osteoarthritis
Brief Title: Nutrition and Movement to Improve Quality of Life With Knee Osteoarthritis
Acronym: NUMOQUA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Pölten University of Applied Sciences (Other)
Collaborators: University of Vienna (Other); Danube University Krems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUMOQUA
Record Dates: First submitted 2023-07-05; First posted 2023-07-21 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Osteo Arthritis Knee
Keywords: Knee; Osteoarthritis; Exercise therapy; Nutrition; Quality of life
MeSH Terms: conditions — Osteoarthritis | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Clinical trial with 2 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training program and nutrition therapy (Experimental): The intervention group receive the GLA:D® training program for 6 weeks and a nutrition therapy for 9 months.
  Interventions: Other: Training program; Other: Nutrition therapy
- Training program (Active Comparator): The control group receive GLA:D® training program for 6 weeks and general information regarding a healthy life style for 9 months.
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — The GLAD training program consists of neuromuscular exercises for the core, the knee and the hip muscles and patient education. The New Nordic Diet is a plant-based nutrition thats aims to reduce systematic low-grad inflammation.
Other: Nutrition therapy — Nutrition therapy based on the New Nordic Diet
  Arms: Training program and nutrition therapy

SUMMARY:
This project aims to evaluate the effects of an evidence-based training program in combination with an antiinflammatory dietetic intervention on quality of life for patients with knee osteoarthritis

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most prevalent arthritic disease worldwide characterized by pain, effusion and stiffness leading to functional decline and reduced quality of life (QL). It has been long considered as a degenerative disease of cartilage resulting from bodily wear and tear that affect the entire joint structure. However, there is accumulating evidence that inflammation plays a key role in the OA pathogenesis. Triggered from tissue damage and by metabolic dysfunction, inflammatory processes within the joint may trigger the development of chronic low-grade inflammation.

Factors that contribute to chronic low-grade inflammation include a nutrient overload, a metabolic surplus, pro-inflammatory cytokines and adipokines. Knee OA is the most common form of OA with prevalence rising with age peaked at around 50 years of age affecting more than 250 million people worldwide. Exercise therapy (ET) is an effective component of early treatment and is therefore recommended as a first line treatment. Good Life with osteoArthritis in Denmark (GLA:D®) represents an evidence-based treatment plan for knee OA and optimizes the implementation of ET. However, ET mainly addresses physical and functional deficits in patients with knee OA, but not the inflammatory processes. Due to the association of chronic low-grad inflammation with dietary patterns, nutrition plays a significant role in inflammation-related diseases. A plant-based, anti-oxidative and anti-inflammatory therapeutic diet helps to improve symptoms leading to improved quality of life. When implementing a therapeutic diet, it should be attractive for patients and regional needs should be considered. This might increase adherence to therapeutic diet and will have an environmental impact - the New Nordic Diet (NND) seems to fulfil these requirements. To our knowledge no study has examined the influence of NND on symptoms and QL in OA. Further, there is a lack of knowledge concerning the impact of exercise therapy AND nutrition therapy on symptoms and QL in patients with knee OA.

Aims

1. To evaluate the effect of a nutrition therapy combined with exercise therapy on QL in patients knee OA
2. To investigate the impact of a nutrition therapy combined with exercise therapy on symptoms, nutrition and inflammation status and joint function in patients with knee OA

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate knee osteoarthritis

Exclusion Criteria:

* Musculosceletal disorders which obviates a participation in the training program
* kognitive deficits
* internal, neurological and mental diseases
* drug and/or alcohol abuse

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-06 (Estimated); Primary Completion 2024-04-02 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (Quality of Life) | 9 Month
  Patient reported outcome measurement, Max: 100, Min: 0, Max is the best that can be achieved

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Sankt Pölten University of Applied Sciences, Sankt Pölten, Lower Austria
  - St. Poelten University of Applied Sciences, Sankt Pölten

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hold E, Chmelar S, Aubram T, Leitner G, Nehrer S, Neubauer O, Wagner KH, Wondrasch B. Nutrition and movement to improve quality of life in patients with knee osteoarthritis: the NUMOQUA study protocol for a randomised controlled trial. Trials. 2024 Apr 9;25(1):245. doi: 10.1186/s13063-024-08048-2. PMID 38594710